CLINICAL TRIAL: NCT04590469
Title: Evidence-Based Supported Digital Intervention for Improving Wellbeing and Health of People Living in Care Homes and Care Home Staff (WHELD) During COVID-19: An RCT to Evaluate COVID-19 Adapted E-WHELD: Benefits and Cost-Effectiveness
Brief Title: Improving Wellbeing and Health for Care Home Residents During COVID-19
Acronym: COVIDWHELD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no longer registered
Sponsor: University of Exeter (Other)
Collaborators: King's College London (Other); London School of Economics and Political Science (Other); University of East Anglia (Other); University of Hull (Other); Alzheimer's Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-21-10
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: 4 month, randomized, parallel group cluster RCT comparing the WHELD nursing home programme with virtual coaching and digital support with treatment as usual
Who Masked: Outcomes Assessor
Masking Description: The intervention is a care home/nursing home training programme/coaching and a digital platform. The research assistants collecting data will do so using virtual platforms and will not be told the randomization of participating care homes. Participating care homes will be told not to disclose treatment allocation, and this will be reinforced by the research assistant at the start of each research assessment to maintain the blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WHELD training/virtual coaching programme supported with digital resources (Experimental): WHELD training/virtual coaching programme supported with digital resources
  Interventions: Other: COVID WHELD
- Treatment as Usual (No Intervention): Usual Best practice

INTERVENTIONS:
Other: COVID WHELD — COVID WHELD is a COVID-19 adapted version of an established nursing home training intervention that confers benefits in well-being and neuropsychiatric symptoms for people with dementia. The adaptations include the development of digital resources to support the programme and virtual coaching.
  Arms: WHELD training/virtual coaching programme supported with digital resources

SUMMARY:
More than 400,000 people in the UK live in care homes. These individuals are particularly vulnerable to COVID-19; many are frail and the majority have concurrent physical health problems and dementia. This group are at the highest risk of becoming severely ill with COVID-19 and are dependent on a stretched care workforce. The isolation, together with the stresses and distressing nature of the current work environment is also likely to have an impact on the mental health and well-being of care staff. It is vital to provide good quality support to enable care staﬀ to remain resilient, and to enable good quality care that maintains the well-being of residents with dementia and reduces emerging neuropsychiatric symptoms in residents without increasing harmful sedative medications.

COVID E-WHELD is based on the optimized WHELD training intervention on successfully completed in randomised clinical trials (RCTs) in 86 care homes, more than 1000 people with dementia. WHELD reduced use of anti-psychotics, improved agitation and overall neuropsychiatric symptoms, improved quality of life and reduced mortality for people with dementia. A digital version of WHELD (eWHELD) with virtual supervision in a further care home RCT including 130 people with dementia has demonstrated beneﬁts for staﬀ carers and improvements in the quality of life of people with dementia, with eWHELD combined with virtual supervision, but not with e-learning alone.

The current project will evaluate a COVID-19 adapted version of eWHELD to address current needs of care homes during the COVID-19 pandemic. This will be undertaken in a 2 arm, 4 month, randomized cluster RCT in 1280 care homes (allowing for 75% drop out with COVID-19 outbreaks) to determine whether COVID-19 adapted eWHELD improves quality of life and mental health for people with dementia in care homes and the mental health of care staff.

DETAILED DESCRIPTION:
COVID E-WHELD: Eﬀectiveness and Cost-Eﬀectiveness

COVID-19 adapted WHELD (with digital resources and virtual coaching) will be compared to usual care in a 4 month randomized, parallel group, cluster RCT with 1280 care homes (allowing for 75% drop out because of COVID-19 outbreaks). Care homes will be randomly assigned to WHELD or treatment as usual in a 1:1 ratio. All care homes receiving treatment as usual will be offered the WHELD intervention after 4 months.

Recruitment will build upon a number of networks and contacts. The investigators already have a network of more than 1300 care homes who would be our ﬁrst point of contact (100 additional care homes from Biomedical Research Centre (BRC) care home network. The investigators have a long established and successful record of recruiting large numbers of care homes to clinical trials (WHELD programme, FITS programme, Pimavanserin programme which involved more than 160 care homes).

Evaluation will be undertaken at baseline, 4 weeks and 4 months post-baseline.

The primary outcome measure will be quality of life in care home residents at 4 months, measured by the DEMQOL proxy, which has shown signiﬁcant beneﬁts in previous WHELD RCTs. The secondary outcomes will include cost-eﬀectiveness (EQ-5D), health utilization, use of sedative medications (anti psychotics, hypnotics), neuropsychiatric symptoms, staﬀ conﬁdence (CODE), staff self-eﬃcacy (SCIDS) and staff mental health (PHQ9) and a COVID-19 tracker.

Process measures collected by coaches will include Goal Attainment,

Assessments will be conducted by telephone or Microsoft Teams, by trained Research Assistants, or with the added option of being collected digitally for staff self-report measures.

Data will also be collected on numbers of remote health and social care (HSC) consultations and on unplanned hospital attendances/admissions (including fall-related injuries). Researchers will also fully cost the COVID eWHELD intervention. To examine the opportunity costs of the intervention, champions will be asked to identify activities that were not undertaken in order to participate and to report any paid and unpaid overtime related to time spent in the champion role. Unit costs will be obtained from nationally applicable sources (PSSRU UC, NHS Reference costs) or calculated anew where necessary.

Key elements of the WHELD intervention include:

* Coaching/training to deliver the WHELD programme which includes person-centred care and person-centred activities and person-centred care plans.
* A COVID-19 speciﬁc resource toolkit - digital bite-sized practical content to stay connected, develop new routines, how to respond to virus-related fear and anxiety
* Facilitated online peer support network for care home managers to share stories and solutions for COVID-19 challenges
* Pooling insights from others to create short, digestible digital resources, such as: checklists, video tips, one-page guides, do's and don'ts, infographics, etc.
* Providing communal, collaborative online group supervision calls, to promote staﬀ well-being and peer-to-peer communities in an online gathering place
* Developing easy reference guides to enable staﬀ to support residents, where appropriate, to use virtual communication tools to stay connected with family and friends
* Providing a series of suggestions, activities, and games all designed to foster connection during a time of isolation

As the intervention is optimized best practice, the researchers would consider this activity as service delivery and not research. The research element is the evaluation of potential benefits for residents and staff, and the evaluation of cost-effectiveness.

Analyses and reporting will follow CONSORT guidance. A full statical analysis plan will be developed during the initial phases of the project and signed oﬀ prior to database lock.

The UK Clinical Research Collaboration (UKCRC)-registered Exeter Clinical Trials Unit will be fully involved in the design, management and governance of the RCT aspects of the trial. The unit will have input into the methodology, provide central trial management/senior oversight, build and test the required data collection systems, undertake randomization, manage the data and ensure a surrounding quality assurance framework.

Care homes will specifically be able to pause participation in the study if there is a COVID-19 outbreak in the care home.

ELIGIBILITY:
Inclusion Criteria:

Care homes which include people with dementia within their client group

All individuals residing in participating care homes who meet diagnostic criteria for dementia and/or score '1' or greater on the Clinical Dementia Rating Scale.

Exclusion Criteria:

Care homes under special measures with the local authority

Residents from whom consent or the advice of a consultee cannot be obtained.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Dementia Quality of Life - DEMQOL proxy | 4 months
  Validated quality of life measure for people with dementia, assessed by informant interview. Minimum score = 32 Maximum score = 128; Higher score denotes better outcome.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory | 4 months
  Standardized assessment of neuropsychiatric symptoms in people with dementia, assessed by informant interview. Minimum score = 0 Maximum score = 144; Higher score denotes worse outcome.
Psychotropic medications | 4 months
  Use of antipsychotic and other psychotropic medications from prescribing charts
Confidence in Dementia (CODE) Scale | 4 months
  Staff confidence measure, self completed questionnaire. Minimum score = 9 Maximum score = 45; Higher score denotes better outcome.
Sense of Competence in Dementia Care Staff (SCIDS) scale | 4 months
  Perceived self efficacy of care staff, self completed questionnaire. Minimum score = 17 Maximum score = 68; Higher score denotes better outcome.
Patient Health Questionnaire (PHQ-9) | 4 months
  Mental Health of care staff, self reported questionnaire. Minimum score = 0 Maximum score = 27; Higher score denotes worse outcome.
EQ5D (Euroquol 5D - 5 dimensions) | 4 months
  A standardized instrument for measuring generic health related quality of life, used for Health economic evaluation. Visual Analogue scale minimum score = 0, maximum score = 100. Higher score denotes better outcome.
Client Service Receipt Inventory | 4 months
  to collect service utilization data for health economics. Assesses cost of service provision; as such no min/max values. Higher value denotes worse cost outcome.

OTHER OUTCOMES:
Goal Attainment Scaling | 4 months
  Ordinal scale to rate progress towards personalized goals for people with dementia as a process outcome. Scale for each goal: Minimum score = 1 Maximum score = 4; Higher score denotes better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Clive Ballard, MD, Principal Investigator — The University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, UK, United Kingdom

REFERENCES:
- [Background] Ballard C, Corbett A, Orrell M, Williams G, Moniz-Cook E, Romeo R, Woods B, Garrod L, Testad I, Woodward-Carlton B, Wenborn J, Knapp M, Fossey J. Impact of person-centred care training and person-centred activities on quality of life, agitation, and antipsychotic use in people with dementia living in nursing homes: A cluster-randomised controlled trial. PLoS Med. 2018 Feb 6;15(2):e1002500. doi: 10.1371/journal.pmed.1002500. eCollection 2018 Feb. PMID 29408901
- [Background] Fossey J, Ballard C, Juszczak E, James I, Alder N, Jacoby R, Howard R. Effect of enhanced psychosocial care on antipsychotic use in nursing home residents with severe dementia: cluster randomised trial. BMJ. 2006 Apr 1;332(7544):756-61. doi: 10.1136/bmj.38782.575868.7C. Epub 2006 Mar 16. PMID 16543297
- [Background] Brooker DJ, Latham I, Evans SC, Jacobson N, Perry W, Bray J, Ballard C, Fossey J, Pickett J. FITS into practice: translating research into practice in reducing the use of anti-psychotic medication for people with dementia living in care homes. Aging Ment Health. 2016 Jul;20(7):709-18. doi: 10.1080/13607863.2015.1063102. Epub 2015 Jul 13. PMID 26167720
- [Background] Ballard C, Banister C, Khan Z, Cummings J, Demos G, Coate B, Youakim JM, Owen R, Stankovic S; ADP Investigators. Evaluation of the safety, tolerability, and efficacy of pimavanserin versus placebo in patients with Alzheimer's disease psychosis: a phase 2, randomised, placebo-controlled, double-blind study. Lancet Neurol. 2018 Mar;17(3):213-222. doi: 10.1016/S1474-4422(18)30039-5. PMID 29452684
- [Background] Smith SC, Lamping DL, Banerjee S, Harwood RH, Foley B, Smith P, Cook JC, Murray J, Prince M, Levin E, Mann A, Knapp M. Development of a new measure of health-related quality of life for people with dementia: DEMQOL. Psychol Med. 2007 May;37(5):737-46. doi: 10.1017/S0033291706009469. Epub 2006 Dec 19. PMID 17176501
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Elvish R, Burrow S, Cawley R, Harney K, Pilling M, Gregory J, Keady J. 'Getting to Know Me': The second phase roll-out of a staff training programme for supporting people with dementia in general hospitals. Dementia (London). 2018 Jan;17(1):96-109. doi: 10.1177/1471301216634926. Epub 2016 Feb 27. PMID 26924840
- [Background] Schepers AK, Orrell M, Shanahan N, Spector A. Sense of competence in dementia care staff (SCIDS) scale: development, reliability, and validity. Int Psychogeriatr. 2012 Jul;24(7):1153-62. doi: 10.1017/S104161021100247X. Epub 2012 Feb 20. PMID 22340666
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Gordon JE, Powell C, Rockwood K. Goal attainment scaling as a measure of clinically important change in nursing-home patients. Age Ageing. 1999 May;28(3):275-81. doi: 10.1093/ageing/28.3.275. PMID 10475864
- [Result] Ballard C, Orrell M, YongZhong S, Moniz-Cook E, Stafford J, Whittaker R, Woods B, Corbett A, Garrod L, Khan Z, Woodward-Carlton B, Wenborn J, Fossey J. Impact of Antipsychotic Review and Nonpharmacological Intervention on Antipsychotic Use, Neuropsychiatric Symptoms, and Mortality in People With Dementia Living in Nursing Homes: A Factorial Cluster-Randomized Controlled Trial by the Well-Being and Health for People With Dementia (WHELD) Program. Am J Psychiatry. 2016 Mar 1;173(3):252-62. doi: 10.1176/appi.ajp.2015.15010130. Epub 2015 Nov 20. PMID 26585409